CLINICAL TRIAL: NCT01088256
Title: Efficacy of Etoricoxib in Patients With Neuropathic Pain With and Without Peripheral Hyperalgesia - A Prove of Concept Trial
Brief Title: Efficacy of Etoricoxib on Peripheral Hyperalgesia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Etoricox09-10; 2009-015496-27 (EudraCT Number)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Causalgia; Polyneuropathy; Postherpetic Neuralgia; Peripheral Nerve Injury; Radiculopathy
Keywords: CRPS; Morbus Sudeck; Causalgia; Etoricoxib; Polyneuropathy; post herpetic neuralgia; peripheral nerve injury; radiculopathy; Nervenverletzung; postherpetische Neuralgie; COX-2-Inhibitor
MeSH Terms: conditions — Causalgia; Polyneuropathies; Neuralgia, Postherpetic; Peripheral Nerve Injuries; Radiculopathy | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- etoricoxib, peripheral hyperalgesia (Active Comparator): 14 patient with neuropathic pain and peripheral hyperalgesia get etoricoxib 90mg for 8 days
  Interventions: Drug: Etoricoxib
- etoricoxib, no peripheral hyperalgesia (Active Comparator): 14 patients with neuropathic pain without peripheral hyperalgesia get etoricoxib 90mg for 8 days
  Interventions: Drug: Etoricoxib
- placebo, peripheral hyperalgesia (Placebo Comparator): 14 patients with neuropathic pain with peripheral hyperalgesia get placebo for 8 days
  Interventions: Drug: placebo
- placebo, no peripheral hyperalgesia (Placebo Comparator): 14 patients with neuropathic pain without peripheral hyperalgesia get placebo for 8 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Etoricoxib — the patients get etoricoxib 90mg for 8 days. They get one pill with 90mg per day
  Other Names: Arcoxia
  Arms: etoricoxib, no peripheral hyperalgesia; etoricoxib, peripheral hyperalgesia
Drug: placebo — patients get one pill of placebo (sugar-pill) per day for 8 days.
  Arms: placebo, no peripheral hyperalgesia; placebo, peripheral hyperalgesia

SUMMARY:
The purpose of the study is to determine the efficacy of etoricoxib on pain patients. The investigators assume that patients with neuropathic pain will have greater pain relief then patients on placebo.

DETAILED DESCRIPTION:
Animal experiments analysing anti-hyperalgesic effects of Coxibs show inconsistent results due to different used dosages and varying different pain models. Theoretical the use of NSAIDs is rational, particularly of Coxibs as a part of the neuropathic pain management. But in the newest topical review, there is no valid information available about the effectiveness of these drugs in human neuropathic pain models or in patients with different underlying mechanism, e.g. with or without hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with
* Persistent moderate or severe pain (> 4 on NRS (1..10)) at rest (average of three daily assessments using a diary for at least two days) .
* Neuropathic pain associated with a clinical and neurologically proven peripheral nerve injury, radiculopathy, postherpetic neuralgia or polyneuropathy or CRPS
* One of the two following QST phenotypes at the baseline assessment:

  * signs of peripheral hyperalgesia (that means, pathological decreased heat pain threshold and/or pathological decreased muscle pain threshold)
  * without signs of peripheral hyperalgesia (no pathological decreased heat - and/or muscle pain threshold)
* Patients of both gender
* Signed consent form
* Patients with the ability to understand and follow the instructions of the doctor

Exclusion Criteria:

* Excluded will be patients Parkinson's disease or a history of cerebral vascular insult or nerve injury.

Excluded will be also all patients with contradictions for the use of Etoricoxib:

* Hypersensitivity to the active substance or to any of the excipients.
* Active peptic ulceration or active gastrointestinal (GI) bleeding.
* Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetyl-salicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors.
* Pregnancy and lactation
* Severe hepatic dysfunction (serum albumin <25 g/l or Child-Pugh score ≥10).
* Estimated renal creatinine clearance <30 ml/min.
* Inflammatory bowel disease.
* Congestive heart failure (NYHA II-IV).
* Patients with hypertension whose blood pressure is persistently elevated above 140/90mmHg and has not been adequately controlled
* Established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease.
* Intake of one of the following drugs (current or in the last 3 days)

  * selective-serotonin-reuptake-inhibitor
  * cetoconazole
  * rifampicin
  * phenytoin
  * carbamazepine
  * dexamethasone or other systemic corticoids
  * traditional nonsteroidal antiphlogistics
  * cyclooxygenase-inhibitors
  * immunosuppressives
  * TNF-α-inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Superior improvement of peripheral hyperalgesia at day six after initiation of Cox-2-inhibiting-medication in comparison to placebo | 12 month

SECONDARY OUTCOMES:
Reduction of the average on-going pain | 12 month
  reduction of the average on-going pain decrease of the neuropathic symptoms intensity (NPSI score) decrease of the patients global impression of change (PGIC) decrease of the frequency and cumulative 7 day dosage of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Dr.med, Study Director — University hospital Bergmannsheil department of pain therapy
Locations (1):
- Bergmannsheil department of pain therapy, Bochum, North Rhine-Westphalia, Germany